CLINICAL TRIAL: NCT02923778
Title: A Phase 2 Study of Talimogene Laherparepvec (T-VEC) and Radiation in Localized Soft Tissue Sarcoma
Brief Title: Talimogene Laherparepvec and Radiation Therapy in Treating Patients With Newly Diagnosed Soft Tissue Sarcoma That Can Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01461; NCI-2016-01461 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1678; 10056 (Other: Dana-Farber - Harvard Cancer Center LAO); 10056 (Other: CTEP); UM1CA186686 (NIH)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Leiomyosarcoma; Liposarcoma; Sarcoma G2; Sarcoma G3; Soft Tissue Sarcoma; Soft Tissue Sarcoma of the Trunk and Extremities; Stage I Soft Tissue Sarcoma AJCC v7; Stage II Soft Tissue Sarcoma AJCC v7; Undifferentiated Pleomorphic Sarcoma
MeSH Terms: conditions — Leiomyosarcoma; Liposarcoma; Sarcoma; Histiocytoma, Malignant Fibrous | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (talimogene laherparepvec, radiation therapy) (Experimental): Patients receive talimogene laherparepvec IT or via intralesional injection at weeks 1, 4, 6 and 8. Beginning 1 week after the start of talimogene laherparepvec, patients undergo radiation therapy on Monday-Friday of weeks 2-6. Patients undergo collection of blood and a tumor biopsy on study and undergo MRI throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Biological: Talimogene Laherparepvec

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Biological: Talimogene Laherparepvec — Given IT or via intralesional injection
  Other Names: ICP34.5-, ICP47-deleted Herpes Simplex Virus 1 (HSV-1) Incorporating the Human GM-CSF Gene; Imlygic; JS1 34.5-hGMCSF 47- pA-; T-VEC

SUMMARY:
This phase II trial studies the side effects of talimogene laherparepvec and radiation therapy and to see how well they work in treating patients with newly diagnosed soft tissue sarcoma that can be removed by surgery (resectable). Biological therapies, such as talimogene laherparepvec, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Radiation therapy uses high energy x-rays, photons. electrons, or protons to kill tumor cells and shrink tumors. Giving talimogene laherparepvec and radiation therapy may work better in treating patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the pathologic complete necrosis rate (the number of patients with >= 95% necrosis divided by the number of evaluable patients) following preoperative treatment with talimogene laherparepvec (T-VEC) in combination with radiation in patients with localized soft tissue sarcoma including a pre-planned interim safety analysis to assess post-surgical wound complications.

SECONDARY OBJECTIVES:

I. To estimate the toxicity of talimogene laherparepvec (T-VEC) in combination with radiation in localized soft tissue sarcomas, during neo-adjuvant treatment and post-surgical resection wound complications.

II. To estimate the rate of radiologic response, prior to surgery, and extent of surgical resection.

III. To estimate time to surgery, time to progression, time to recurrence, and death.

CORRELATIVE OBJECTIVES:

I. To characterize the clinical outcomes within three distinct histologic subtypes: liposarcoma (excluding myxoid liposarcoma), leiomyosarcoma and undifferentiated pleomorphic sarcoma.

II. To characterize the percentage of tumor necrosis in treated tumors. III. To assess if the combination of preoperative talimogene laherparepvec (T-VEC) with radiation will increase the expression of PD-L1 in soft tissue sarcomas.

IV. To assess the impact of preoperative talimogene laherparepvec (T-VEC) with radiation on the tumor infiltrating and circulating immune cells in patients with soft tissue sarcomas.

OUTLINE:

Patients receive talimogene laherparepvec intratumorally (IT) or via intralesional injection at weeks 1, 4, 6 and 8. Beginning 1 week after the start of talimogene laherparepvec, patients undergo radiation therapy on Monday-Friday of weeks 2-6. Patients undergo collection of blood and a tumor biopsy on study and undergo magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then every year for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years

  * Note: Because no dosing or adverse event data are currently available on the use of talimogene laherparepvec (T-VEC) in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Newly diagnosed and a histopathologically confirmed potentially resectable soft tissue sarcoma of the extremity or trunk of the following subtypes:

  * Cohort 1: liposarcoma (excluding myxoid liposarcoma)
  * Cohort 2: leiomyosarcoma
  * Cohort 3: undifferentiated pleomorphic sarcoma (UPS) (malignant fibrous histiosarcoma [MFH])
  * NOTE: If local pathology report is suggestive of or suspicious for UPS, study chair and study pathologists may review for eligibility determination.
  * NOTE: Sites permissible for biopsy include

    * Extremities: upper (including shoulder) and lower (including hip)
    * Trunk: Body wall
* Patients must have a histologically determined grade 2 or 3 tumor by the French Federation of Cancer Centers Sarcoma Group (FNCLCC) sarcoma grading system
* Patients must have localized disease with a primary tumor > 5 cm by MRI or computed tomography (CT) scan
* Patients must have a primary tumor that is determined by multidisciplinary team (medical oncology, orthopedic/surgical oncology, and radiation oncology) to require radiation therapy for optimal management prior to surgical resection
* Patients must have a sarcoma in the extremity or trunk in location, which is accessible to direct or ultrasound guided injections
* Karnofsky performance score >= 70
* Absolute neutrophil count (ANC) >= 1500/uL
* Absolute lymphocyte count (ALC) >= 800/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN
* Calculated creatinine clearance > 70 mL/min/1.73 m^2
* Patient must have a life expectancy of at least 3 months with appropriate therapy
* Patients must agree to use contraception during study treatment and for 4 months after the end of treatment

  * NOTE: Talimogene laherparepvec (T-VEC), as well as other therapeutic agents used in this trial, may cause fetal harm when administered to a pregnant woman; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation, and for four months after the last dose of the drug; women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to registration and agree to use effective contraception throughout the treatment period and for 4 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to provide mandatory blood and tissue samples for correlative studies and central pathology confirmation of surgical specimens collected during study participation
* Willingness to provide a tissue sample that is mandatory at the time of surgery (if applicable) and the determination of the primary objective of the study

Exclusion Criteria:

* Patients with localized sarcomas that are not of the extremity or trunk wall (including head/neck, retroperitoneum, visceral organs, peritoneum, pelvis within the confines of the bony pelvis, and tumors arising in bone)
* Patients who have had prior treatment with anti-PD1 or anti-CTLA4 therapy
* Patients with grade 1 non-rhabdomyosarcoma soft tissue sarcomas (NRSTS) tumors of any size are not eligible
* Patients with evidence of active bleeding or bleeding diathesis will be excluded (patients with excess of 2.5 mL of hemoptysis are not eligible)
* Patients requiring any therapeutic anticoagulation
* Patients must have had no prior radiotherapy to tumor-involved sites
* Patients with gross total resection of the primary tumor or who have developed tumor recurrence after gross total tumor resection prior to enrollment are not eligible
* History of serious or non-healing wound, ulcer, or bone fracture
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1)
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of talimogene laherparepvec (T-VEC) and during the study
* Previous treatment with talimogene laherparepvec (T-VEC) or any other oncolytic virus
* Patients with metastatic disease
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to talimogene laherparepvec (T-VEC) or any of its components
* History or evidence of active autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other); or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) within 2 months of enrollment; (replacement therapy [e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency] is not considered a form of systemic treatment for autoimmune disease)

  * Evidence of clinically significant immunosuppression such as

    * Primary immunodeficiency state such as severe combined immunodeficiency disease
    * Concurrent opportunistic infection
    * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 2 months prior to enrollment
* Active herpetic skin lesions or prior complications of herpetic infection (e.g., herpetic keratitis or encephalitis)
* Viral infections requiring intermittent or chronic systemic (intravenous or oral) treatment with an anti-herpetic drug, other than intermittent topical use (e.g., acyclovir)
* Other viral infections

  * Known to have acute or chronic active hepatitis B or hepatitis C infection
  * Known to have human immunodeficiency virus (HIV) infection
  * Prior therapy with viral-based tumor vaccine
  * Received live vaccine within 28 days prior to enrollment
* Patients who are unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for herpes simplex virus (HSV)-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or children under the age of 1 year, during talimogene laherparepvec (T-VEC) treatment and through 30 days after the last dose of talimogene laherparepvec (T-VEC)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant, breastfeeding or plan to become pregnant

  * NOTE: Although no effects on embryo-fetal development have been observed in animal studies, adequate and well-controlled studies with talimogene laherparepvec (T-VEC) have not been conducted in pregnant women; therefore, sexually active patients and their partners must be willing to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation, and for four months after the last dose of T-VEC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (CR) rate | Up to 5 years
  Will be defined as >= 95% of tumor having necrosis. The estimated pathologic CR rate and a 95% confidence interval will be reported.
Incidence of post-surgical wound complications | Up to 4 months post-surgery
  Evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Incidence of toxicities of T-VEC in combination with radiation therapy | Up to 5 years
  Will be evaluated according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Summary statistics and frequency tables will be used to describe the distributions of the observed adverse events occurring pre-surgery and following surgery. All patients having initiated study treatment will be considered evaluable for toxicity analysis.
Rate of radiologic response | Up to 5 years
  Will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Estimates and confidence intervals will be used to summarize the observed rate of radiologic response.
Rate of surgical response | Up to 5 years
  Will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Estimates and confidence intervals will be used to summarize the observed rate of surgical response.
Time to surgery | From registration date until surgery, assessed up to 5 years
  Will be estimated using Kaplan-Meier methodology.
Time to progression | From registration date until disease progression, assessed up to 5 years
  Will be estimated using Kaplan-Meier methodology.
Time to recurrence | From registration date until disease recurrence, assessed up to 5 years
  Will be estimated using Kaplan-Meier methodology in only those patients having achieved a complete surgical resection.
Time to death | From registration date until death, assessed up to 5 years
  Will be estimated using Kaplan-Meier methodology.

OTHER OUTCOMES:
Clinical outcomes within liposarcoma, leiomyosarcoma, and undifferentiated pleomorphic sarcoma | Up to 5 years
Percentage of tumor necrosis in treated tumors | Up to 5 years
  Summary statistics and frequency tables will be used to describe tumor necrosis. T-tests, logistic regression, and non-parametric methods, if required, may be used.
Change in PD-L1 expression | Baseline to time of surgery
Change in tumor infiltrating and circulating immune cells | Baseline to time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Steven I Robinson, Principal Investigator — Mayo Clinic Cancer Center LAO
Locations (17):
- United States (16):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Goff PH, Riolobos L, LaFleur BJ, Spraker MB, Seo YD, Smythe KS, Campbell JS, Pierce RH, Zhang Y, He Q, Kim EY, Schaub SK, Kane GM, Mantilla JG, Chen EY, Ricciotti R, Thompson MJ, Cranmer LD, Wagner MJ, Loggers ET, Jones RL, Murphy E, Blumenschein WM, McClanahan TK, Earls J, Flanagan KC, LaFranzo NA, Kim TS, Pollack SM. Neoadjuvant Therapy Induces a Potent Immune Response to Sarcoma, Dominated by Myeloid and B Cells. Clin Cancer Res. 2022 Apr 14;28(8):1701-1711. doi: 10.1158/1078-0432.CCR-21-4239. PMID 35115306